CLINICAL TRIAL: NCT03369561
Title: Comparison Between Right and Left Ventricular Systolic Dysfunction as a Risk Factors for AKI in Critical Care Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Noura gamal, principle Investigator, Assiut University
Other Study IDs: CBRALVSDASRFFAKICCP
Record Dates: First submitted 2017-11-25; First posted 2017-12-12 (Actual); Last update posted 2017-12-12 (Actual); Status verified 2017-12

CONDITIONS: Acute Kidney Injury (Nontraumatic)
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- normal cardiac patient: Full history and clinical examination ECG on the left and right side Echocardiography and measurement of both left and right ventricular functions Laboratory investigation including cardiac enzymes, CK, CK MB, and cardiac troponin I.
  Serum urea and creatinine and the calculated e GFR
  Interventions: Diagnostic Test: Serum urea and creatinine and the calculated e GFR

INTERVENTIONS:
Diagnostic Test: Serum urea and creatinine and the calculated e GFR — The primary outcome will be AKI during the 1st 7 days of ICU care, as defined by an increase of ≥ 0.3 mg/dl in serum creatinine within 48 hours of ICU admission, an increase of ≥ 50% within 7 days of ICU admission, or acute dialysis

SUMMARY:
The cardio renal syndrome generally focuses on left ventricular function, and the importance of the right ventricle as a determinant of renal function is described less frequently. Although the risk of AKI is similar for patients with isolated LVD and isolated RVD, the severity of AKI and the associated risk of hospital mortality is highest among those with isolated RVD.

DETAILED DESCRIPTION:
The right ventricle seems to affect renal function through different mechanisms, including Venous Congestion, tricuspid regurgitation, And potential inhibitory effect on left ventricular function The most important mechanism is venous congestion, a manifestation of sodium avidity and fluid expansion, as Directly increasing renal venous pressure causes sodium retention, lowers urinary output, and decreases glomerular filtration and widely thought to explain AKI Venous pressure is directly associated with renal dysfunction, independently of ventricular function, and admission peripheral edema is associated with greater risk of AKI. Such awareness of a primary role of renal venous congestion reshapes our understanding of renal function as not simply a reflection of arterial perfusion, but rather a balance between arterial supply and venous drainage.

.

ELIGIBILITY:
Inclusion Criteria:

* cardiac patient

Exclusion Criteria:

* ESRD pt CKD Cirrhotic patients AKI due to post renal cause

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All pt admitted to ICU with Lt , Rt or Bi ventricular dysfunction That develops AKI
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2018-01-01 (Estimated); Primary Completion 2019-01-01 (Estimated); Study Completion 2020-03-01 (Estimated)

PRIMARY OUTCOMES:
AKI during the 1st 7 days of ICU care, | One year
  defined by an increase of ≥ 0.3 mg/dl in serum creatinine within 48 hours of ICU admission, an increase of ≥ 50% within 7 days of ICU admission, or acute dialysis, in keeping with the Kidney Disease Improving Global Outcomes guidelines.

CONTACTS AND LOCATIONS:
Overall Officials: Ashraf M El-Shazly, Prof, Study Chair — Assiut
Locations (1):
- Assiut University Hospital, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Legrand M, Mebazaa A, Ronco C, Januzzi JL Jr. When cardiac failure, kidney dysfunction, and kidney injury intersect in acute conditions: the case of cardiorenal syndrome. Crit Care Med. 2014 Sep;42(9):2109-17. doi: 10.1097/CCM.0000000000000404. PMID 24810531
- [Background] Liang KV, Williams AW, Greene EL, Redfield MM. Acute decompensated heart failure and the cardiorenal syndrome. Crit Care Med. 2008 Jan;36(1 Suppl):S75-88. doi: 10.1097/01.CCM.0000296270.41256.5C. PMID 18158481
- [Background] F Gnanaraj J, von Haehling S, Anker SD, Raj DS, Radhakrishnan J. The relevance of congestion in the cardio-renal syndrome. Kidney Int. 2013 Mar;83(3):384-91. doi: 10.1038/ki.2012.406. Epub 2012 Dec 19. PMID 23254894
- [Background] Palevsky PM, Liu KD, Brophy PD, Chawla LS, Parikh CR, Thakar CV, Tolwani AJ, Waikar SS, Weisbord SD. KDOQI US commentary on the 2012 KDIGO clinical practice guideline for acute kidney injury. Am J Kidney Dis. 2013 May;61(5):649-72. doi: 10.1053/j.ajkd.2013.02.349. Epub 2013 Mar 15. PMID 23499048
- [Background] van Walraven C, Austin PC, Jennings A, Quan H, Forster AJ. A modification of the Elixhauser comorbidity measures into a point system for hospital death using administrative data. Med Care. 2009 Jun;47(6):626-33. doi: 10.1097/MLR.0b013e31819432e5. PMID 19433995
- [Background] Gutacker N, Bloor K, Cookson R. Comparing the performance of the Charlson/Deyo and Elixhauser comorbidity measures across five European countries and three conditions. Eur J Public Health. 2015 Feb;25 Suppl 1:15-20. doi: 10.1093/eurpub/cku221. PMID 25690125